CLINICAL TRIAL: NCT04568330
Title: Re-validating Prophylactic Efficacy of Urea-based Cream on Sorafenib-induced Hand-foot Skin Reaction in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Prevention of Hand-foot Skin Reaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Jiin Ger, MD, Taipei Veterans General Hospital, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013-11-009
Record Dates: First submitted 2020-08-29; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: hand-foot skin reaction; side effect of sorafenib; symptom related to target therapy; efficacy of urea-based cream; symptom management
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Best support care (BSC) (Other): Interventions for comparison group (group C) who received BSC alone were (1) informed of potential presentations of HFSR, (2) asked for wearing waterproof gloves before execute household or work with water, (3) provided the method of contacting with healthcare specialists for confirming early diagnosis of HFSR, and (4) asked for self-report when they occurred symptoms of HFSR.
  Interventions: Other: best support care
- BSC plus moisture cream (Experimental): The A group with BCS plus moisturizing cream received the interventions as the comparison group, was given the moisturizing cream (dimethicone, fragrance free, Aveeno, United States) for 9 times and was instructed how to use the cream. The education of usage included (1) using the cream twice a day from 3 days before starting sorafenib and each week post starting sorafenib, (2) scooping out nut-sized cream with a unique spoon each time, (3) gently applied the cream evenly on symmetrical palms below wrists and symmetrical soles below ankles each time, (4) wore unique cotton gloves immediately after the appalment of cream for 30 minutes each time.
  Interventions: Other: moisture cream
- 10% urea-based cream (Active Comparator): The B group with BCS plus 10% urea-based cream had the similar interventions as the A group with BCS plus moisturizing cream except being given the cream container with different component (10% urea; Sipharr, Taiwan). The outlook of the containers with the two kinds of cream was the same. All the cream looks white and grey.
  Interventions: Other: 10% urea-based cream

INTERVENTIONS:
Other: best support care — Best support care
  Arms: Best support care (BSC)
Other: moisture cream — BSC plus moisture cream
  Arms: BSC plus moisture cream
Other: 10% urea-based cream — BSC plus 10% urea-based cream.
  Arms: 10% urea-based cream

SUMMARY:
Sorafenib-induced hand-foot skin reaction (HFSR) is a dose-dependent side effect in patients with advance hepatocellular carcinoma (HCC). The appropriate prophylactic dose of urea-based cream and comparison of its effectiveness with other creams remain unclear. The aim of this study was re-validating the prophylactic HFSR incidence density and cutaneous wetness of 10% urea-based cream on sorafenib-induced HFSR in patients with advanced HCC.

DETAILED DESCRIPTION:
Methods

Patients

This study population consisted of patients with (1) HCC by proof of pathology, (2) presence of tumor thrombus in the main trunk of the portal vein or the first-order branches of the portal vein with minimal ascetics or with no ascetics by abdominal CT scan, (3) Child-Pugh liver function class A, (4) planning to receive oral sorafenib 400 mg twice per day, (5) age of 20 or more years old, and (6) able to communication in Chinese, Taiwanese or Hakka. Patients with (1) encephalopathy, psychosis, cognition impairment, blindness or hearing impairment, (2) allergic history to urea, (3) present ulceration, blisters, infective problems on the palms or soles, or (4) previous surgery, systematic chemotherapy or frequent radial ablation were excluded.

Research procedure

This is a randomized double-blind experiment study. Sample size was estimated by the G. power software version 3.1, which was set with logistic regression, odds ratio: 3.8, and power: 0.80. The estimated sample size should be 125 at least. This study, there was recruited 129 patients (43 patients in each groups). All eligible patients were recruited from Taipei Veterans General Hospital between January 1st and December 31th, 2014. They were randomly assigned in a ratio of 1:1:1 to treat with best supportive care plus moisturizing cream (A group), BSC plus 10% urea-based cream (B group) and BSC alone (group C which is comparison group),by method of EXCEL random sampling. A case manager recruited the eligible patients who also conducted informed consent and patient education. A research employee had responsibilities to record patients' demographic data, provide non-label cream and check previous container of the cream that should be exhausted. A medical oncologist or a nurse had responsibilities to assess patients' severity of HFSR and cutaneous wetness. The assessment was done on 3 days before starting sorafenib treatment and each 7 days after the starting, total 9 times. Creams were provided after the assessment. When patients developed HFSR, they will be referred to receive the most appropriate management.

Interventions

Interventions for group C (comparison group) who received BSC alone were (1) informed of potential presentations of HFSR, (2) asked for wearing waterproof gloves before execute household or work with water, (3) provided the method of contacting with healthcare specialists for confirming early diagnosis of HFSR, and (4) asked for self-report when they occurred symptoms of HFSR. The A group with BCS plus moisturizing cream received the interventions as the comparison group, was given the moisturizing cream (dimethicone, fragrance free, Aveeno, United States) for 9 times and was instructed how to use the cream. The education of usage included (1) using the cream twice a day from 3 days before starting sorafenib and each week post starting sorafenib, (2) scooping out nut-sized cream with a unique spoon each time, (3) gently applied the cream evenly on symmetrical palms below wrists and symmetrical soles below ankles each time, (4) wore unique cotton gloves immediately after the appalment of cream for 30 minutes each time. A B group with BCS plus 10% urea-based cream had the similar interventions as the A group with BCS plus moisturizing cream except being given the cream container with different component (10% urea; Sipharr, Taiwan). The outlook of the containers with the two kinds of cream was the same. All the cream looks white and grey.

Outcomes and assessment

Data of con founders and two end-points, incidence density of HFSR and cutaneous wetness, were collected. The con-founders included gender, age, numbers of chronic illnesses, numbers of metastatic regions as well as levels of white count, hemoglobin, bleeding time, liver enzymes, albumin and electrolyte.

The grades of HFSR were assessed by NCI-CTCAE version 4, which was developed by Dueck et al. This is an available psychometric patient-reported instrument. Body water with 33% or less meant dry skin, 34% to 37% meant mild dry skin, 38% to 42% meant general status, 43% to 46/% was mild moisty skin and 47% or more presented moisty skin. When using the scanner, examiners had to confirm whether it tied to fix on the skin.

Ethical considerations

This study was approved by the Institution Review Board of the Taipei Veterans General Hospital (2013-13-009B). Informed consent was obtained from all patients by a case manager on 3 days before starting sorafenib. Patients were explained the study protocol and were educated self-care skills by the case manager. All of them were well aware that their rights will be protected, the risk of participation will be limited to the lowest and most suitable management will be arranged when they developed sorafenib-induced HFSR.

ELIGIBILITY:
Inclusion Criteria:

* HCC by proof of pathology
* Presence of tumor thrombus in the main trunk of the portal vein or the first-order branches of the portal vein with minimal ascetics or with no ascetics by abdominal CT scan
* Child-Pugh liver function class A
* Planning to receive oral sorafenib 400 mg twice per day
* Age of 20 or more years old
* Able to communication in Chinese, Taiwanese or Hakka

Exclusion Criteria:

* Encephalopathy, psychosis, cognition impairment, blindness or hearing impairment
* Allergic history to urea
* Present ulceration, blisters, infective problems on the palms or soles
* Previous surgery, systematic chemotherapy or frequent radial ablation

Ages: 54 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-03-21 (Actual); Primary Completion 2015-11-11 (Actual); Study Completion 2015-12-11 (Actual)

PRIMARY OUTCOMES:
Scale | three days before taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 3.0

SECONDARY OUTCOMES:
Scale | 1 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)

OTHER OUTCOMES:
Scale | 2 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Scale | 3 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Scale | 4 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Scale | 5 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Scale | 6 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Scale | 7 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Scale | 8 week after taking Sorafenib
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Benson AB 3rd, Abrams TA, Ben-Josef E, Bloomston PM, Botha JF, Clary BM, Covey A, Curley SA, D'Angelica MI, Davila R, Ensminger WD, Gibbs JF, Laheru D, Malafa MP, Marrero J, Meranze SG, Mulvihill SJ, Park JO, Posey JA, Sachdev J, Salem R, Sigurdson ER, Sofocleous C, Vauthey JN, Venook AP, Goff LW, Yen Y, Zhu AX. NCCN clinical practice guidelines in oncology: hepatobiliary cancers. J Natl Compr Canc Netw. 2009 Apr;7(4):350-91. doi: 10.6004/jnccn.2009.0027. No abstract available. PMID 19406039
- [Background] Kao PH, Cen JS, Chung WH. Cutaneous adverse events of targeted anticancer therapy: a review of common clinical manifestations and management. J Cancer Res Pract. 2015; 2(4): 271-284.
- [Background] Wood LS, Lemont H, Jatoi A. Practical considerations in the management of hand-foot skin reaction caused by multikinase inhibitors. Commun Oncol .2010; 7: 23-39
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Result] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Result] Cubero DIG, Abdalla BMZ, Schoueri J, Lopes FI, Turke KC, Guzman J, Del Giglio A, Filho CDSM, Salzano V, Fabra DG. Cutaneous side effects of molecularly targeted therapies for the treatment of solid tumors. Drugs Context. 2018 Jul 17;7:212516. doi: 10.7573/dic.212516. eCollection 2018. PMID 30038659
- [Result] Lipworth AD, Robert C, Zhu AX. Hand-foot syndrome (hand-foot skin reaction, palmar-plantar erythrodysesthesia): focus on sorafenib and sunitinib. Oncology. 2009;77(5):257-71. doi: 10.1159/000258880. Epub 2009 Nov 16. PMID 19923864
- [Result] Massey PR, Okman JS, Wilkerson J, Cowen EW. Tyrosine kinase inhibitors directed against the vascular endothelial growth factor receptor (VEGFR) have distinct cutaneous toxicity profiles: a meta-analysis and review of the literature. Support Care Cancer. 2015 Jun;23(6):1827-35. doi: 10.1007/s00520-014-2520-9. Epub 2014 Dec 5. PMID 25471178
- [Result] Chang WT, Lu SN, Rau KM, Huang CS, Lee KT. Increased cumulative doses and appearance of hand-foot skin reaction prolonged progression free survival in sorafenib-treated advanced hepatocellular carcinoma patients. Kaohsiung J Med Sci. 2018 Jul;34(7):391-399. doi: 10.1016/j.kjms.2018.03.006. Epub 2018 Apr 4. PMID 30063012
- [Result] Macdonald JB, Macdonald B, Golitz LE, LoRusso P, Sekulic A. Cutaneous adverse effects of targeted therapies: Part I: Inhibitors of the cellular membrane. J Am Acad Dermatol. 2015 Feb;72(2):203-18; quiz 219-20. doi: 10.1016/j.jaad.2014.07.032. PMID 25592338
- [Result] Manchen E, Robert C, Porta C. Management of tyrosine kinase inhibitor-induced hand-foot skin reaction: viewpoints from the medical oncologist, dermatologist, and oncology nurse. J Support Oncol. 2011 Jan-Feb;9(1):13-23. doi: 10.1016/j.suponc.2010.12.007. PMID 21465734
- [Result] Ren Z, Zhu K, Kang H, Lu M, Qu Z, Lu L, Song T, Zhou W, Wang H, Yang W, Wang X, Yang Y, Shi L, Bai Y, Guo X, Ye SL. Randomized controlled trial of the prophylactic effect of urea-based cream on sorafenib-associated hand-foot skin reactions in patients with advanced hepatocellular carcinoma. J Clin Oncol. 2015 Mar 10;33(8):894-900. doi: 10.1200/JCO.2013.52.9651. Epub 2015 Feb 9. PMID 25667293
- [Result] Negri FV, Porta C. Urea-Based Cream to Prevent Sorafenib-Induced Hand-and-Foot Skin Reaction: Which Evidence? J Clin Oncol. 2015 Oct 1;33(28):3219-20. doi: 10.1200/JCO.2015.61.6417. Epub 2015 Jul 27. No abstract available. PMID 26215963
- [Result] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Result] Dueck AC, Mendoza TR, Mitchell SA, Reeve BB, Castro KM, Rogak LJ, Atkinson TM, Bennett AV, Denicoff AM, O'Mara AM, Li Y, Clauser SB, Bryant DM, Bearden JD 3rd, Gillis TA, Harness JK, Siegel RD, Paul DB, Cleeland CS, Schrag D, Sloan JA, Abernethy AP, Bruner DW, Minasian LM, Basch E; National Cancer Institute PRO-CTCAE Study Group. Validity and Reliability of the US National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). JAMA Oncol. 2015 Nov;1(8):1051-9. doi: 10.1001/jamaoncol.2015.2639. PMID 26270597
- [Result] Piccoli A, Rossi B, Pillon L, Bucciante G. A new method for monitoring body fluid variation by bioimpedance analysis: the RXc graph. Kidney Int. 1994 Aug;46(2):534-9. doi: 10.1038/ki.1994.305. No abstract available. PMID 7967368
- [Result] Shinohara N, Nonomura N, Eto M, Kimura G, Minami H, Tokunaga S, Naito S. A randomized multicenter phase II trial on the efficacy of a hydrocolloid dressing containing ceramide with a low-friction external surface for hand-foot skin reaction caused by sorafenib in patients with renal cell carcinoma. Ann Oncol. 2014 Feb;25(2):472-6. doi: 10.1093/annonc/mdt541. Epub 2013 Dec 18. PMID 24351402
- [Result] Barton-Burke M, Ciccolini K, Mekas M, Burke S. Dermatologic Reactions to Targeted Therapy: A Focus on Epidermal Growth Factor Receptor Inhibitors and Nursing Care. Nurs Clin North Am. 2017 Mar;52(1):83-113. doi: 10.1016/j.cnur.2016.11.005. PMID 28189168
- [Derived] Lien RY, Tung HH, Wu SL, Hu SH, Lu LC, Lu SF. Validation of the prophylactic efficacy of urea-based creams on sorafenib-induced hand-foot skin reaction in patients with advanced hepatocellular carcinoma: A randomised experiment study. Cancer Rep (Hoboken). 2022 Jul;5(7):e1532. doi: 10.1002/cnr2.1532. Epub 2021 Dec 14. PMID 34910380